CLINICAL TRIAL: NCT01628887
Title: Feasibility of a Supportive Education Program for Latina Breast Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Proposal will not be submitted and low accrual.
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12175
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Cancer Survivor; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (BBCEI) (Experimental): Participants undergo 2 tailored BBCEI sessions within 1 month. At the beginning of the first session the research nurse will present the participants with a list of common physical and social concerns. The participant will then be asked to identify 3 topics that she wants to discuss. The research nurse will discuss with the participant any relevant supportive care resources and make the appropriate referrals. At the second session the focus of the BBCEI will be on psychological and spiritual well-being.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Undergo Bilingual Breast Cancer Educational Intervention

SUMMARY:
This clinical trial studies a supportive education program for Latina breast cancer survivors. The Bilingual Breast Cancer Education Intervention (BBCEI) may help Latina breast cancer survivors know what to expect after completing breast cancer treatment and prepare them to cope with cancer related survivorship issues

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Describe the feasibility of implementing the BBCEI. II. Describe the cultural and linguistic appropriateness of the BBCEI. III. Determine topics requiring further emphasis in the BBCEI. IV. Identify ways to enhance program content, format, and materials. OUTLINE: Participants undergo 2 tailored BBCEI sessions within 1 month. At the beginning of the first session the research nurse will present the participants with a list of common physical and social concerns. The participant will then be asked to identify 3 topics that she wants to discuss. The research nurse will discuss with the participant any relevant supportive care resources and make the appropriate referrals. At the second session the focus of the BBCEI will be on psychological and spiritual well-being.

ELIGIBILITY:
The population will consist of Latinas with breast cancer who have completed primary cancer treatment. A total of 10 subjects will be accrued.

Inclusion Criteria:

* Diagnosis of Stage I, II or III.
* Self-identification as Hispanic/Latina.
* Able to read and understand English or Spanish to participate in the education sessions.
* Ability to read and/or understand the study protocol requirements, and provide written informed consent
* Subjects maybe be on hormonal therapy after treatment for initial breast cancer.

Exclusion Criteria:

* Actively receiving treatment with surgery, radiation therapy, or chemotherapy.
* Patients who have recurrence, metastasis, or a second primary cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of implementation of a Bilingual Breast Cancer Education Intervention (BBCEI) | 2 months after completion of the educational session
  A semi-structured interview guide will be used to describe participant satisfaction with the BBCEI. It allows the patient to describe in their own words whether the BBCEI was effective for their QOL concerns, helpfulness of intervention content, describe the cultural and linguistic appropriateness and identify ways to enhance program content, format and materials.
Determine the cultural and linguistic appropriateness of the BBCEI | 2 months after completion of the educational session
  A semi-structured interview guide will be used to describe participant satisfaction with the BBCEI. It allows the patient to describe in their own words whether the BBCEI was effective for their QOL concerns, helpfulness of intervention content, describe the cultural and linguistic appropriateness and identify ways to enhance program content, format and materials
Determine topics requiring further emphasis in the BBCEI | 2 months after completion of the educational session
  A semi-structured interview guide will be used to describe participant satisfaction with the BBCEI. It allows the patient to describe in their own words whether the BBCEI was effective for their QOL concerns, helpfulness of intervention content, describe the cultural and linguistic appropriateness and identify ways to enhance program content, format and materials
Determine ways to enhance program content, format and materials | 2 months after completion of the educational session
  A semi-structured interview guide will be used to describe participant satisfaction with the BBCEI. It allows the patient to describe in their own words whether the BBCEI was effective for their QOL concerns, helpfulness of intervention content, describe the cultural and linguistic appropriateness and identify ways to enhance program content, format and materials

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Juarez, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States